CLINICAL TRIAL: NCT04999501
Title: Comparison of the Benefits of Prolonged Resistance-type Exercise Training in the Older Population Aged 65-75 y Versus 85 y and Over
Brief Title: Resistance-type Exercise Training in the Older Population
Acronym: RETO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Gabriel Nasri Marzuca-Nassr, Professor, Universidad de La Frontera
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FONDECYT 11180949
Record Dates: First submitted 2021-07-26; First posted 2021-08-11 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Aged, 80 and Over; Resistance Training
Keywords: oldest old; exercise; muscle mass; strength; functional capacity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 65 - 75 years (Experimental): All volunteers aged 65 - 75 will be subjected to 12 weeks of full body resistance exercise training (3 times per week).
  Interventions: Other: Prolonged resistance-type exercise training
- 85 years and over (Experimental): All volunteers over the age of 85 will be subjected to 12 weeks of full body resistance exercise training (3 times per week).
  Interventions: Other: Prolonged resistance-type exercise training

INTERVENTIONS:
Other: Prolonged resistance-type exercise training — All volunteers will be subjected to 12 weeks of whole-body resistance-type exercise training (3x/wk).

SUMMARY:
Background: Aging is associated with muscle mass and strength loss and "oldest" old people (≥85 y) are at a far greater risk of developing sarcopenia. Training increases muscle mass and strength in a variety of populations, yet the efficacy has not been clearly defined for individuals in the fourth age (≥80 y).

Hypothesis: The following hypotheses will be investigated:

* Twelve weeks of progressive resistance-type exercise training increases muscle mass and strength in young old (65-75 y) and oldest old (85 y and over) subjects.
* The training-induced increase in muscle mass and strength is relatively greater in young old subjects when compared to oldest old subjects.

Goals: The primary aim of this study is to compare the effect of resistance-type exercise training on skeletal muscle mass (i.e. quadriceps cross-sectional area and whole body lean mass) in young old and oldest old subjects.

Specific goals

* Determine whether resistance-type exercise training can increase muscle mass and muscle strength in young old and oldest old subjects.
* Determine whether resistance-type exercise training can improve physical performance in young old and oldest old subjects.
* Identify whether inflammatory markers (i.e., TNFα, IL-4, IL-6, IL-10, IL-13) are up- or down-regulated in young old and oldest old subjects before and after resistance-type exercise training.

Methodology:

Study design Sixty older females and males (young old group: n=30, 65-75 y; oldest old group: n=30, 85 y and over) will be included in this prospective clinical trial. All volunteers will be subjected to 12 weeks of whole-body resistance-type exercise training (3x/wk). Before, and after 6 and 12 weeks of training, a computed tomography (CT) scan of the upper leg will be performed to assess quadriceps cross sectional area. On those days, fasting blood samples will be obtained and whole-body dual energy x-ray absorptiometry (DEXA) scan will also be performed. Maximal strength will be determined by 1-repetition maximum (1RM) and physical functioning by the short physical performance battery (SPPB) at the same time points.

DETAILED DESCRIPTION:
Background: Aging is associated with muscle mass and strength loss and "oldest" old people (≥85 y) are at a far greater risk of developing sarcopenia. Training increases muscle mass and strength in a variety of populations, yet the efficacy has not been clearly defined for individuals in the fourth age (≥80 y). A better understanding of the skeletal muscle adaptive response to resistance-type exercise training with advanced age will provide a strong basis to develop and implement care programs within our rapidly aging population, in which the "oldest" old represent the fastest growing group.

Hypothesis: The following hypotheses will be investigated:

* Twelve weeks of progressive resistance-type exercise training increases muscle mass and strength in young old (65-75 y) and oldest old (85 y and over) subjects.
* The training-induced increase in muscle mass and strength is relatively greater in young old subjects when compared to oldest old subjects.

Goals: The primary aim of this study is to compare the effect of resistance-type exercise training on skeletal muscle mass (i.e. quadriceps cross-sectional area and whole body lean mass) in young old and oldest old subjects.

Specific goals

* Determine whether resistance-type exercise training can increase muscle mass and muscle strength in young old and oldest old subjects.
* Determine whether resistance-type exercise training can improve physical performance in young old and oldest old subjects.
* Identify whether inflammatory markers (i.e., TNFα, IL-4, IL-6, IL-10, IL-13) are up- or down-regulated in young old and oldest old subjects before and after resistance-type exercise training.

Methodology:

Study design Sixty older females and males (young old group: n=30, 65-75 y; oldest old group: n=30, 85 y and over) will be included in this prospective clinical trial. All volunteers will be subjected to 12 weeks of whole-body resistance-type exercise training (3x/wk). Before, and after 6 and 12 weeks of training, a computed tomography (CT) scan of the upper leg will be performed to assess quadriceps cross sectional area. On those days, fasting blood samples will be obtained and whole-body dual energy x-ray absorptiometry (DEXA) scan will also be performed. Maximal strength will be determined by 1-repetition maximum (1RM) and physical functioning by the short physical performance battery (SPPB) at the same time points.

Study parameters/endpoints

* The main study endpoint is the increase in quadriceps cross-sectional area as assessed via CT scan.
* Secondary endpoints include: Whole-body and segmental body composition (i.e., lean mass, fat mass, bone mineral content; DEXA scan); Maximal strength assessment (1RM); Hand grip strength; Short physical performance battery (SPPB); Inflammatory and molecular markers (blood samples analysis).
* Other study parameters include: Age, body weight, body height, body mass index (BMI), lipid profile, glucose, and insulin.

Expected results:

The impact of resistance-type exercise training to increase muscle mass and strength in the oldest old population remains unclear. With the proposed project, we expect that resistance-type exercise training will increase muscle mass and strength, although the impact will be relatively lower in the oldest old group when compared with a group of young old individuals. The potential findings will define the efficacy of resistance-type exercise training to increase muscle mass and strength in individuals with advancing age. Better maintenance, or even an increase in muscle mass and strength increases independence, prolonging good health, recovery from disease and illness, and ultimately decreases burden on healthcare systems. This information will have a beneficial impact in the exercise physiology and aging areas for future interventions at the local, regional, national and international levels.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 65-75 and 85 and more years.
* 18.5 < BMI < 30 kg/m2.
* Older people that are still "community-dwelling", i.e., not living in a nursing-home or elderly-home.

Exclusion Criteria:

* Performing regular resistance training (2 or more times per week, carrying out progressive training) in the previous 6 months.
* Cardiovascular diseases that are contradictory for physical activity (not included controlled Hypertension).
* All co-morbidities interacting with mobility and muscle metabolism of the body and that do not allow to (safely) perform the resistance-type exercise program (e.g. debilitating arthritis, spasticity/rigidity, all neurological disorders and paralysis).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change in skeletal muscle mass (measured via Computed tomography (CT) scan) after prolonged resistance-type exercise training | Before, and after 6 and 12 weeks of training
  Cross-sectional area of the quadriceps and L3 region via single-slice CT scan

SECONDARY OUTCOMES:
Change in lean tissue (measured via Dual Energy X-ray Absorptiometry (DEXA) scan) after prolonged resistance-type exercise training | Before, and after 6 and 12 weeks of training
  Measurement of Whole Body Composition via DEXA
Change in arms and legs strength (measured via 1-Repetition Maximum (1RM) testing) after prolonged resistance-type exercise training | Before, and after 6 and 12 weeks of training
  Maximal strength assessment via 1RM testing of horizontal row, lat pull down, chest press, leg press, and leg extension)
Change in hand grip strength (measured via JAMAR handheld dynamometer) after prolonged resistance-type exercise training | Before, and after 6 and 12 weeks of training
  Maximal strength assessment via 1RM testing of JAMAR handheld dynamometer.
Change in physical performance (measured via Short physical performance battery (SPPB)) after prolonged resistance-type exercise training | Before, and after 6 and 12 weeks of training
  Measurement of physical performance via SPPB
Change in Inflammatory markers via ELISA after prolonged resistance-type exercise training | Before, and after 6 and 12 weeks of training,
  Measurement in blood samples via ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Faculty of Medicine, Universidad de La Frontera. Temuco, Chile, Temuco, Chile

IPD SHARING:
Plan to Share IPD: Undecided